CLINICAL TRIAL: NCT06901882
Title: Evaluation of the Effectiveness of Training in Basic and Assisted Communication Techniques for Intensive Care Nurses: A Quasi-experimental Study
Brief Title: Nursing Interventions in Communication for the Critically Ill Patient: CONECTEM Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Marta Prats Arimon, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: reference PR(AG)120/2019
Record Dates: First submitted 2025-03-03; First posted 2025-03-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Nurse-patient Communication
Keywords: augmentative and alternative communication; training program; psicoemotional effects; nurse-patient relationship
MeSH Terms: conditions — Critical Illness | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design with two groups, Intervention group and control group with a pre-post test model.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: CONECTEM, Communication based in BCS (basic communication skills) and AAC ( aumentative alternative communicatiton)
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: CONECTEM, Communication based in BCS (basic communication skills) and AAC ( aumentative alternative communicatiton) — It consists of applying basic and assisted communication techniques, already validated by experts (Happ, et al., 2008) to the critical patient admitted to the ICU. The intervention is divided into 3 strategies according to the level of patient awareness. Each strategy presents both verbal and non-verbal communication skills
  Estratègia 3. Glasgow (≤8). Very ill patient, with indications for intubation, sedation and analgesia. We will basically use non-verbal communication, taking into account all external factors that may predispose to a change in the patient's condition.
  Modulate your voice, speak softly and slowly, respecting an atmosphere of silence, without intense lights or loud noises. Adjust the temperature of the ICU according to the needs of the patient.
  Achieve a relaxing atmosphere, playing calm music during the journey.Make comforting movements for the patient, avoiding abruptness and trying to establish non-verbal communication.
  Arms: Intervention group

SUMMARY:
The aim of this quasi-experimental study is to find out whether the effectiveness of a communication intervention based on basic and assisted communication techniques improves the psycho-emotional effects of critical patients admitted to an ICU. The nurses' knowledge of BCS and CAA and their usefulness in daily practice will also be investigated. The main questions to be answered are:

Does effective communication based on BCS and CAA reduce pain, anxiety and stressful impact of the critically ill in the ICU? Do nurses who apply these communication techniques believe that they are useful in their daily practice?

The researchers will compare the communicative intervention called 'CONECTEM' with the usual nurse-patient communication process to observe whether CBT and CCT are effective in decreasing the psycho-emotional effects of these patients.

Participants will:

Participants will be classified into 3 groups according to the Glasgow Coma Scale, for each group different communicative strategies based on scientific literature will be applied. In each strategy, different theories such as Carkkuff, Light and different levels of support (no technology, low technology) will be used. The intervention has a minimum duration of 15 minutes and before and after the 3 variables studied will be evaluated. The intervention will be carried out during the first 72 hours after admission.

Prior to the intervention, a formal training in BCS and ACC will be given to the nurses who will then apply the intervention.

DETAILED DESCRIPTION:
CONECTEM Training Programme: This programme is aimed at nurses in the intensive care unit who will carry out communicative intervention with critically ill patients. It consists of 4 blocks, with a theoretical part and a practical part, in which the nurses acquire knowledge, skills and attitudes related to basic and assisted communication with the critically ill. The theoretical part is based on the theories of R Carkuff (2008)(1), and the Augmentative Assistive Communication model (2,3), and the practical part consists of a series of verbal and non-verbal communication exercises, and of experiencing communication simulations with the critically ill patient using the appropriate techniques and material.

The training programme also explains how the CONECTEM Communicative Intervention is carried out in Phase II. This training programme consists of two 2-hour sessions and will be evaluated by means of a theoretical-practical test to see if the nurses who carry out the intervention in phase II are able to carry it out.

CONECTEM Communication Intervention: This consists of applying basic and assisted communication techniques, already validated by experts (4) to the critical patient admitted to the ICU. The intervention is divided into 3 strategies according to the level of patient awareness. Each strategy presents both verbal and non-verbal communication skills and appropriate material for patients with communication difficulties (physical or cognitive). Each strategy includes details of the specific communication techniques to be used by the therapists and a description of how they are to be used.

Procedure and data collection Phase I: Procedure for the selection of participants. Depending on the participation of the ICU nurses of the study hospital who meet the inclusion/exclusion criteria, they will be given a folder made up of: a) full information and informed consent, b) a form to collect socio-demographic variables c) forms to collect the variables of knowledge on communication with the critically ill. Of all the nurses participating in this phase, 16 nurses will be selected by agreement to participate in phase II, who will be assigned to the control group or the intervention group. Training in the CONECTEM programme will be given to the 8 nurses who form part of the intervention group. Once the training has been completed, a test will be used to assess whether the nurses are able to carry out the CONECTEM Communicative Intervention with critical patients . The questionnaire on perceived satisfaction with the training programme will also be completed . All these data will be collected by the research team.

Phase II:

The selection of patients will be by consecutive cases, as they enter the ICU. Participants will have to comply with the specified inclusion and exclusion criteria and will have to sign the informed consent form (either on their own or delegated). The data collection will be carried out by the IG and CG nurses. The IG nurses will be given a folder that will include: a) a form of socio-demographic and health variables of the patient , b) the detailed CONECTEM Communicative Intervention, c) the scales for the evaluation of the psycho-emotional variables studied and d) a questionnaire on the usefulness of the CONECTEM training programme . The CG nurses will be given a folder with a) a form of socio-demographic and health variables of the patient and b) scales for the evaluation of the psycho-emotional effects. Data collection will be carried out twice a year until the patient is discharged from the ICU. In the IC, the nurse will collect the data pre-post CONECTEM communicative intervention, which lasts a minimum of 15 minutes. The nurses of the CG will collect the pre-post data pre-post nurse-patient interaction on a regular basis.

Annex 4

1. Training in basic and assisted communication techniques (CONECTEM)

   The theoretical part; Based on three theories on nurse-patient communication:

   Theory of 'Helping Human Relationships'(1): Based on a model of effective communication where 2 basic sets of skills are defined in the communicative activity: the initiation dimension and the response dimension. The nurse and the patient carry out a joint reflexive process in order to be successful in the therapeutic relationship.

   Theory of 'Interpersonal Relations in Nursing' (5): Based on therapeutic communication between nurse and patient, the foundations of which are: transparency, respect, dialogue and non-verbal communication. It proposes an integral vision of the infernal cures where effective communication is the essence.

   'Augmentative Assistive Communication (AAC) (2,3): A communication system for people with temporary or permanent communication difficulties and/or limitations who are unable to express and/or understand themselves verbally and/or in writing in their daily lives.It consists of classifying the real communicative needs of the disabled into 4 functions: expression of needs or desires, development of the close social circle, exchange of information and social behaviour routines.

   In this theoretical part, the psycho-emotional effects of the critically ill are also described, the particularities of the Care Unit are emphasised and the communicative intervention that will be carried out during phase II is explained (strategies, variables and measuring instruments).

   The practical part consists of exercises in trusting others, non-verbal communication exercises, emotional work and the application, in a fictitious situation, of basic and assisted communication techniques.

   Training objectives - To understand the importance of communication in critical illness.
   * Know how to recognise psychoemotional disorders (pain, stress and anxiety).
   * Learn new communication techniques with critically ill people who present communication difficulties of comprehension and/or expression.
   * To learn techniques for communicating with unconscious patients.
   * Improve basic communication skills. Assessment of the training
   * Theoretical-practical exam to see if nurses achieve the established objectives and can therefore participate in phase II of the project.
   * The perceived satisfaction of the training in basic and assisted communication techniques will be evaluated once it has been completed.
   * The perception of the usefulness of the training in basic and assisted communication techniques will be assessed 3 months after starting the CONECTEM communication intervention.

   Material and methodology
   * The course will last 2 hours and will be held in ten different times so that all nurses can attend.
   * Power Point support and audiovisual media such as some videos and images. Work in small groups to discuss the examples presented and emotional work will be done. Role-palying for the simulation of cases.
   * Non-verbal communication and confidence exercises with peers will be carried out using materials such as a snot-brush, a paper clipboard, cardboard and coloured paper.
2. CONECTEM Communicative Intervention It consists of applying a series of communicative strategies, previously validated in the literature (3,4). The intervention classifies the communicative techniques into three groups according to the patient's state of consciousness. Each group of strategies involves a level of verbal and non-verbal communication.

Strategy 1. Glasgow 15. The patient is conscious and oriented, has no difficulty in understanding or expressing him/herself in order to communicate.

We will use verbal and non-verbal communication. This strategy will be based on Carkhuff's 'Helping human Relation-ships theory', which shows the basis for achieving a positive relationship between the patient and the nurse by means of two key dimensions: The response dimension (empathy, respect, clarity in expression) and the initiative dimension (showing authenticity, open-mindedness/non-judgement, confronting one's own feelings, being concrete) (1).

Description and authors of the communicative actions of Strategy 1 of CONECTEM intervention STRATEGY/AUTHOR ACTION TO BE CARRIED OUT Gain attention and visual contact (2) Make sure that the patient and the nurse are focused on each other, both with their gaze and with the messages.

Confirm all the patient's messages (3).Validate that the message has been understood by repeating the message or what has been understood about the message.

Make pauses (2). Allowing more time between communication exchanges facilitates the patient's thought process.

Yes/no sentence ending strategy (3). Making sentences or questions with yes/no at the end alerts the patient that he/she will have to choose an option.

Clarity of expression (1). Clarify and verify the perception of the message. Paraphrasing, short and simple sentences.

Empathy and active listening (1). Understanding the patient's concerns, desires, worries, etc... helps the flow of communication.

Respect (1). Accepting others as they are without judging them. Assertiveness (1). Modulate the language, tone of voice, intentionality of the emitter allowing feedback with the other.

Own elaboration, based on the authors of the table. Strategy 2. Glasgow (14-9). Conscious, disoriented person with difficulties in communicating due to gravity.

We will use verbal and non-verbal communication. If the patient has the ability to speak, we will use Strategy 1 plus Strategy 2. (1,3) We can see the communicative strategies in the following table.

Description and authors of the communicative actions of Strategy 2 of the CONECTEM intervention.

STRATEGY/AUTHOR ACTION TO BE CARRIED OUT Concreteness and precision in language (1). Use short phrases or simple sentences with yes/no at the end to make it easier for the patient to understand.

Establish a clear yes/no signal e.g.: moure el cap amunt/avall = yes. (2,3). Ensure that the yes/no signal can be carried out and remembered by the patient and understood by others.

Patient gestures or international signs - dictionary (4,6). Perform international signs to establish feedback with the patient.

Communicative assistance with drawings (3,4). Use the banners where there are a series of drawings with the patient's needs. The patient must point out the need and this will be repeated aloud by the nurse.

Own elaboration based on the authors of the table. b-1 Signs of the universal dictionary (4)

b-2 Patient Emotion Indicator Panel (4)

b-3 Patient needs indicator panel. (4)

Estratègia 3. Glasgow (≤8). Very ill patient, with indications for intubation, sedation and analgesia. We will basically use non-verbal communication, taking into account all external factors that may predispose to a change in the patient's condition. The communication strategies described in the following table can be observed.

. Description and authors of the communicative actions of Strategy 3 of the CONECTEM intervention.

STRATEGY/AUTHOR ACTION TO BE PERFORMED Facial expression and motor movements (3).Observe facial gestures and movements, especially those of the extremities. These will be the most reliable indicators of comfort/uncomfort, pain/non-pain expression, stress/non-stress...

Alteration of physical signs (7). Controlling changes in HR, BP, RR, sweating Tonality of voice and calm environment (4).

Musique (8,9). Modulate your voice, speak softly and slowly, respecting an atmosphere of silence, without intense lights or loud noises. Adjust the temperature of the ICU according to the needs of the patient.

Achieve a relaxing atmosphere, playing calm music during the journey (10). Make comforting movements for the patient, avoiding abruptness and trying to establish non-verbal communication.

ELIGIBILITY:
Inclusion Criteria:

* Critical patients admitted to the ICU's of the Hospital Vall d'Hebron who accepted to participate in the study on their own volition or by delegation of the family member, previously informed in writing.

Exclusion Criteria:

* Patients who do not understand Catalan or Spanish, critically ill patients admitted to the ICU for less than 24 hours and/or diagnosed with a psychiatric disorder prior to admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Level of pain | VAS: Pre-post intervention (0 -30 minutes), Pre-post Nursing care (0-30 minutes). Glasgow >9. BPS: Pre-post intervention (0 -30 min), Pre-post Nursing care (0-30 min). Glasgow <9
  VAS Visual Analògic scale for mesuring pain for responsable patients Consists of a 10-centimetre horizontal line, at the ends of which are the extreme expressions of a symptom. On the left is the absence of the symptom and on the right the highest intensity. The patient is asked to indicate on the line what intensity of the symptom is present.
  Behabiour Pain Scale for unresponsable patients. It is divided into 5 items that assess facial expression and motor movements. Each item is scored from 0 to 2 in a graded manner. The sum of all the items gives a score that indicates the state of the pain according to whether it is mild, moderate or intense, with 0 being painless and 12 being the maximum intensity of pain.
Level of anxiety for responsable patients | Pre post intervention 0-30 minutes, pre post nursing usual care 0-30 minutes. Glasgow >9
  the STAI Scale short version (Perpiña-Galvañ 2013), which consists of 6 items that are divided into 2 categories; present anxiety and absent anxiety.
Level of sedation and agitation | Pre-post intervention 0 -30 minutes , Pre post nursing usual care 0-30 minutes ( glasgow <9)
  RASS (sedation and agitation scale), which consists of 9 items ranging from -5 to 4 and assesses the agitation and degree of sedation of the patient under mechanical ventilation. From -5 to -1 the patient is sedated, the lower the number the less negative the degree of sedation will be. 0 is alert and calm, and from 1 to 4 the patient is agitated, anxious with possible acute psychological disorders. The higher the value, the more intense the scale, with 1 being restless and 4 combative
level of post-traumatic stress symptoms | Pre post intervention 0-30 minutes , pre post nursing usual care 0-30 minutes. Gasgow >9
  Stressor Impact Scale (EIE) (Badia-Castelló 2006), which is made up of 15 items: 6 measure intrusiveness, 8 avoidance and 1 hyperarousal. The score for each item is measured from 0 to 5, being 0 never, 1 sometimes, 3 often, 5 frequently. From the total score it is established that PTE LLEU<8,5 PTE moderate 8,5-19 and PTE severe >19
level of consciousness | Baseline
  Glasgow Coma Scale (Tesdale 1974). The scale is divided into three independently scorable groups that evaluate eye opening over 4 points, verbal response over 5 points and motor response over 6 points, with the maximum score (conscious and oriented) being 15 and the minimum 3.

SECONDARY OUTCOMES:
perception of the usefulness of the CONECTEM intervention | 3 month post data collection
  - The variable perception of the usefulness of the CONECTEM intervention will be assessed on the basis of a questionnaire made by the research team consisting of 8 items. It is measured on a Likert-type scale ranging from not at all (1), a little (2), often (3), quite a lot (4), a lot (5).

OTHER OUTCOMES:
Sex | Baseline
  % de males and females using a socialdemographic questionnaire Sex
  1. Male
  2. Female
Age in years | Baseline
  Age in whole numbers
educational Level | Baseline
  % and frecuencies of educational level by socio-demographic questionnaire
  1. Primary school studies (school-leaving certificate, ESO)
  2. Intermediate vocational training cycle
  3. Batxillerat, Cicles formatius de grau superior (baccalaureate, higher vocational training courses)
  4. University degree
  5. Doctoral studies
  6. No studies
  7. Other studies (non-regulated studies) say which ones
Marital status | Baseline
  % and frecuencies of marital status by socio-demographic questionnaire
  1. Single
  2. Married
  3. Divorced
  4. Widowed
  5. Unmarried partner
Origin/nationality | Baseline
  % and frecuencies origin/nationality ofpatients using socio-demographic questionnaire
  1. Place of birth:
  2. Province:
  3. Country:
Employment situation | Baseline
  % and frecuencies employment situation of patients using socio-demographic questionnaire
  1. Permanent job
  2. Interim
  3. Substitute
  4. Unemployed
  5. Retirement
TYPE OF PATHOLOGY | Baseline
  % and frecuencies of patient's pathology using a questionnaire
  1. Cardiac
  2. Respiratory
  3. Neurological
  4. Traumatic
  5. Metabolic
  6. Other (ex medical) enter what
patient on mechanical ventilation | Baseline
  % and frecuencies of patient on mechanical ventilation using a questionnaire
  1. yes
  2. no
communicative strategy used | Pre-intervention
  Strategy n 1 (Glasgow 15) Strategy n 2 (Glasgow 14-9) Strategy n 3 (Glasgow < 9)
Hearing impairment | Baseline
  It is used to assess whether the patient is hearing impaired using a questionnaire. (% and frequencies)
  1. yes
  2. no
  3. need a device holder
Visual Impairment | Baseline
  It is used to assess whether the patient is visual impaired using a questionnaire (% and frequencies)
  1. Yes
  2. No
  3. wears glasses
Motor impairment | Baseline
  It is used to assess whether the patient is motor impaired using a questionnaire (% and frequencies)
  1. Generalised fatigue
  2. Hemiparesis D
  3. Hemiparesis E
  4. Facial paralysis
  5. EEII (paraplegia)
  6. Tetraplegia
  7. Dysarthria
  8. None
Cognitive impairment | Baseline
  It is used to assess whether the patient cognitive impaired using a questionnaire (% and frequencies)
  1. Attention deficit
  2. Comprehension deficit
  3. Expressive aphasia
  4. Comprehension aphasia
  5. Memory loss
  6. Illusory memory (hallucinations, distortion of reality)
  7. None

CONTACTS AND LOCATIONS:
Overall Officials: Marta Prats-Arimon, PHD, Principal Investigator — University of Barcelona
Locations (1):
- University of Barcelona, L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradt J, Dileo C. Music interventions for mechanically ventilated patients. Cochrane Database Syst Rev. 2014;2014(12):CD006902. doi: 10.1002/14651858.CD006902.pub3. Epub 2014 Dec 9. PMID 25490233
- [Background] Beukelman DR, Fager S, Ball L, Dietz A. AAC for adults with acquired neurological conditions: a review. Augment Altern Commun. 2007 Sep;23(3):230-42. doi: 10.1080/07434610701553668. PMID 17701742
- [Background] Puntillo KA, Max A, Timsit JF, Vignoud L, Chanques G, Robleda G, Roche-Campo F, Mancebo J, Divatia JV, Soares M, Ionescu DC, Grintescu IM, Vasiliu IL, Maggiore SM, Rusinova K, Owczuk R, Egerod I, Papathanassoglou ED, Kyranou M, Joynt GM, Burghi G, Freebairn RC, Ho KM, Kaarlola A, Gerritsen RT, Kesecioglu J, Sulaj MM, Norrenberg M, Benoit DD, Seha MS, Hennein A, Periera FJ, Benbenishty JS, Abroug F, Aquilina A, Monte JR, An Y, Azoulay E. Determinants of procedural pain intensity in the intensive care unit. The Europain(R) study. Am J Respir Crit Care Med. 2014 Jan 1;189(1):39-47. doi: 10.1164/rccm.201306-1174OC. PMID 24262016
- [Background] Happ MB, Baumann BM, Sawicki J, Tate JA, George EL, Barnato AE. SPEACS-2: intensive care unit "communication rounds" with speech language pathology. Geriatr Nurs. 2010 May-Jun;31(3):170-7. doi: 10.1016/j.gerinurse.2010.03.004. Epub 2010 May 10. PMID 20525521
- [Background] Gastmans C. Interpersonal relations in nursing: a philosophical-ethical analysis of the work of Hildegard E. Peplau. J Adv Nurs. 1998 Dec;28(6):1312-9. doi: 10.1046/j.1365-2648.1998.00840.x. PMID 9888377
- [Background] Light J. Communication is the essence of human life: Reflections on communicative competence. AAC Augment Altern Commun. 1997;13(2):61-70
- [Background] Happ MB, Sereika S, Garrett K, Tate J. Use of the quasi-experimental sequential cohort design in the Study of Patient-Nurse Effectiveness with Assisted Communication Strategies (SPEACS). Contemp Clin Trials. 2008 Sep;29(5):801-8. doi: 10.1016/j.cct.2008.05.010. Epub 2008 Jun 7. PMID 18585481
- [Background] Carkhuff R. The Art of Helping. 9a ed. HRD Press I, editor. Amherst; U.S; Canada: Possibilities Publishing; Inc; 2009. 302 p.
- [Background] Arimon MP, Llobet MP, Roldan-Merino J, Moreno-Arroyo C, Blanco MAH, Lluch-Canut T. A Communicative Intervention to Improve the Psychoemotional State of Critical Care Patients Transported by Ambulance. Am J Crit Care. 2021 Jan 1;30(1):45-54. doi: 10.4037/ajcc2021619. PMID 33385200
- See also: This programme consists of providing nurses with the tools and resources they need to communicate effectively with critically ill patients — https://diposit.ub.edu/dspace/handle/2445/125752